CLINICAL TRIAL: NCT07372781
Title: Clinical Study on the Early Bactericidal Activity of Contezolid Against Mycobacterium Abscessus Disease
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Chest Hospital (Other)
Responsible Party: Principal Investigator, Nie WenJuan, chief physician, Beijing Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCP-TB-2024-11-15
Record Dates: First submitted 2025-01-28; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Monotherapy; Mycobacterium Abscessus Infection
Keywords: early bactericidal activity; colony forming units; Time To Positivity; Mycobacterium abscessus
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous | interventions — contezolid; Oxazolidinones; Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contezolid group (Experimental): Contezolid 800mg twice daily for 14 days. To enroll 12 patients with Mycobacterium abscessus infections, who will receive continuous administration of contezolid for 14 days. Sputum samples will be collected for colony forming units counting and Time To Positivity observation to evaluate the Early Bactericidal Activity.
  Interventions: Drug: Contezolid
- Linezolid group (Active Comparator): Linezolid 600mg once daily for 14 days. To enroll 12 patients with Mycobacterium abscessus infections, who will receive continuous administration of linezolid for 14 days. Sputum samples will be collected for colony forming units counting and Time To Positivity observation to evaluate the Early Bactericidal Activity.
  Interventions: Drug: linezolid

INTERVENTIONS:
Drug: Contezolid — Patients with Mycobacterium abscessus infections were enrolled and treated with a 14-day monotherapy of contezolid for anti-Mycobacterium abscessus therapy, through analysis and comparison of colony forming units and Time To Positivity in sputum cultures.
  Other Names: Oxazolidinone
  Arms: Contezolid group
Drug: linezolid — Patients with Mycobacterium abscessus infections were enrolled and treated with a 14-day monotherapy of linezolid for anti-Mycobacterium abscessus therapy, through analysis and comparison of colony forming units and Time To Positivity in sputum cultures.
  Other Names: Oxazolidinone
  Arms: Linezolid group

SUMMARY:
This study is a single-center, randomized, controlled, open-label clinical trial designed to assess the early bactericidal activity of a single agent, contezolid, in patients with Mycobacterium abscessus infections. Patients were administered contezolid monotherapy for 14 days specifically targeting Mycobacterium abscessus, and were compared to a control group receiving linezolid, a classic anti-Mycobacterium abscessus drug. The comparison was conducted through the analysis of colony forming units counts and Time To Positivity in sputum cultures. By evaluating the impact of contezolid monotherapy on the bacterial load in the sputum of patients with Mycobacterium abscessus infections, this study aimed to assess the early bactericidal activity of contezolid, thereby providing a basis for the selection of new therapeutic options for the treatment of patients with Mycobacterium abscessus infections.

DETAILED DESCRIPTION:
As one of the drugs for treating Mycobacterium abscessus infections, linezolid is effective but its use is limited in anti-Mycobacterium abscessus treatment regimens due to the high incidence of adverse reactions associated with long-term use. Contezolid, a new drug developed in China, belongs to the oxazolidinone class of drugs and shares a similar antibacterial spectrum with linezolid, while exhibiting a significantly better safety profile. This study is a single-center, randomized, controlled, open-label clinical trial designed to evaluate the early bactericidal activity. It enrolls patients with Mycobacterium abscessus disease and administers a 14-day monotherapy of contezolid for the treatment of the disease. The study compares contezolid with linezolid, a classic anti-Mycobacterium abscessus drug, by analyzing colony forming units and Time To Positivity in sputum cultures. By assessing the impact of contezolid monotherapy on the bacterial load in the sputum of patients with Mycobacterium abscessus disease, the study evaluates the early bactericidal activity of contezolid, providing a basis for the selection of new therapeutic options for the treatment of Mycobacterium abscessus disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 18 and 65 years old;
* Weight ranging from 40 kg to 90 kg;
* At least one positive sputum culture for Mycobacterium abscessus within 6 months prior to screening, and one positive sputum culture for Mycobacterium abscessus with molecular species identification during the screening period within 1 month prior to the study;
* Voluntary participation in this study and signing of the informed consent form; (5) Male and female participants must use effective contraception during the study and for 1 month after the study ends.

Exclusion Criteria:

* Patients who have been on long-term corticosteroid therapy or taking immunosuppressants within 90 days prior to screening;
* Pregnant women, postpartum women, and lactating patients;
* Patients with a history of bedaquiline allergy or known hypersensitivity, or a history of severe adverse reactions;
* Patients with evidence of bedaquiline resistance;
* Patients deemed unsuitable for participation in this study by the investigator's assessment;
* Patients whom the investigator believes participation in this study would harm their health, or who are unlikely to comply with the scheduled visits and assessments as outlined in the protocol, and therefore are not suitable for participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time To Positivity in sputum cultures | 14 days
  With a 14-day monotherapy of contezolid for anti-Mycobacterium abscessus therapy, then were compared with a control group receiving linezolid, a classic anti-Mycobacterium abscessus drug, through analysis and comparison of Time To Positivity in sputum cultures.

CONTACTS AND LOCATIONS:
Overall Officials: Wenjuan Nie, Director, Study Director — Beijing Tuberculosis & Thoracic Tumor Research Institute Beijing Chest Hospital affiliated to Capital Medical University
Locations (1):
- Beijing chest hospital affiliated to Capital medical university, Beijing Tuberculosis & Thoracic Tumor Research Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
In our hospital, the investigators are not allowed to casually publish participants' information and hospital data on the website.